CLINICAL TRIAL: NCT02663154
Title: Aromatherapy for Postoperative Nausea and Vomiting in Children: A Single Blind Randomized Clinical Trial
Brief Title: Aromatherapy for Postoperative Nausea and Vomiting in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stuart Wright (Other)
Collaborators: Soothing Scents, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Stuart Wright, Assistant Professor, Dept of Pediatric Anesthesia, IWK Health Centre, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1016941
Record Dates: First submitted 2015-12-23; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Aromatherapy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aromatherapy (Experimental): Aromatherapy inhaler (QueaseEASE, Soothing Scents Inc, Enterprise, AL) applied to nauseous post surgical paediatric patients in the postanesthetic care unit
  Interventions: Drug: Aromatherapy inhaler
- Placebo (Placebo Comparator): Saline inhaler applied to nauseous post surgical paediatric patients in the postanesthetic care unit
  Interventions: Drug: Saline inhaler

INTERVENTIONS:
Drug: Aromatherapy inhaler — Inhalation of commercial essential oil preparation (QueaseEASE) delivered in the commercial inhaler package in postanesthetic care unit after surgery in paediatric patients complaining of nausea
  Other Names: QueaseEASE (Soothing Scents, Inc, Enterprise, AL)
  Arms: Aromatherapy
Drug: Saline inhaler — Inhaler is similar in design and function as the intervention inhaler only with saline rather than essential oils. Inhaler provided by the manufacturer QueaseEASE (Soothing Scents, Inc, Enterprise, AL)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most common postoperative complications of general anesthesia in pediatrics. Pediatric rates of nausea and vomiting are approximately double those of adult patients. Aromatherapy has recently been shown to reduce PONV in adults, but the effect in paediatric patients is unknown. The goal of this study is to determine the feasibility of a large-scale study in the paediatric population.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of the most common postoperative complications of general anesthesia occurring after up to 40% of general anesthetics. PONV is an unpleasant experience and can result in secondary complications including wound dehiscence, electrolyte abnormalities and aspiration pneumonia. PONV often causes delayed stays in the postanesthesia care unit and delayed hospital discharge.

The mechanism of PONV is poorly understood. Given the multifactorial nature of nausea and vomiting, standard pharmacological therapy approaches the problem from various pathways. Methods that include antihistaminic therapies such as dimenhydrinate (gravol), antiserotonergic medications such as ondansetron (Zofran) and glucocorticoids (dexamethasone), have been used effectively in different surgical settings to address PONV. They do not work however, without occasional significant side effects such as urinary retention, blurred vision, increased infection rates, headaches and constipation. Given that pharmacological interventions for PONV are not universally effective and have accompanying side effects, there has been recent interest in additional complementary interventions.

Aromatherapy has been used to treat nausea from motion sickness, pregnancy, cancer and pain. In postoperative adults, a recent large adequately powered randomized control trial found aromatherapy resulted in a significant risk reduction of nausea (0.37) when compared with saline. Given the encouraging results of the first adequately powered adult study, the goal is to determine whether PONV is reduced by aromatherapy in the pediatric population. Thus, the primary aim of this study is to determine if aromatherapy is more effective than placebo in the treatment of postoperative nausea in children as a complementary treatment to current postoperative practices.

This research is important as it is the first study to assesses whether aromatherapy can be useful in postoperative nausea treatment for children. The implications of this study could mean an improvement in the health care experience of children who have nausea postoperation and potentially a reduction in rescue antinausea drug use in this population in the future.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I or II
* absence of neurodevelopment disorders
* patient having elective day surgery

Exclusion Criteria:

* family or patient refusal
* allergy or sensitivity to aromatherapy oils
* inability to smell in the postoperative period

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reduction in postoperative nausea and vomiting score | 2 hours postoperative in the post anesthetic care unit
  A validated nausea scale called the Baxter Animated Retching Faces (BARF) scale will be administered to the patient in the postanesthetic care unit.
  Upon arrival in the postanesthesia care unit the research assistant will assess for nausea using the BARF scale at 15-minute intervals. If the patient reports a BARF scale of 4 or greater, they will be entered into the study and randomized to a placebo or aromatherapy inhaler.
  The primary outcome is defined as a two-point reduction in the BARF scale. This has been shown to be a clinically significant effect in the paediatric nausea literature.

SECONDARY OUTCOMES:
Total number of patients who used antiemetics | 2 hours post-operatively
  The use of antiemetic by patients enrolled in the study at any time in the 2 hour post-operative period will be recorded as yes or no and expressed as the number of patients who needed antiemetics compared to the total number of patients in the intervention arm.
Total number of patients with emesis | 2 hours post-operatively
  The total number of patients who vomit in the 2 hour post-operative period.
Total number of patients who continue to use the inhaler | 2 hours post-operatively
  Total number of patients who continue use of the study inhaler post first dose of aromatherapy or placebo.
Reduction in Baxter Animated Retching Faces (BARF) scale magnitude | 2 hours post-operatively
  Patients enrolled in the study in the postanesthetic recovery unit will be administered the BARF scale post-intervention with the placebo or aromatherapy inhaler. The magnitude of the reduction in the BARF scale will be recorded for each subject. The net reduction number in the BARF scale will be averaged and expressed as the number with confidence intervals for each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Wright, MD, Principal Investigator — IWK Health Centre

REFERENCES:
- [Derived] Kiberd MB, Clarke SK, Chorney J, d'Eon B, Wright S. Aromatherapy for the treatment of PONV in children: a pilot RCT. BMC Complement Altern Med. 2016 Nov 9;16(1):450. doi: 10.1186/s12906-016-1441-1. PMID 27829428